CLINICAL TRIAL: NCT01777789
Title: The Role of Mid-Life Adiposity in Functional Brain Connectivity
Status: Terminated | Type: Observational
Why Stopped: This is a basic research study with no clinical data to report
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: PRO16109
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Alzheimer's Disease
Keywords: fMRI; Dementia; Alzheimer's disease; functional neuroimaging; Memory
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood draw
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to use functional MRI (fMRI) to measure brain connectivity in middle-aged individuals with different levels of body fat. The ultimate goal of this research is to develop an early diagnostic tool for Alzheimer's disease.

DETAILED DESCRIPTION:
Participants will have one visit for:

* Blood draw
* Body composition scan
* Cognitive screen
* Neurological exam
* MRI scan

The visit will take approximately 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* 45-65 years of age
* Normal memory
* Right-handed
* General good physical health

Exclusion Criteria:

* History of stroke or neurological disease
* Seizures or head injury with loss of consciousness within the last five years
* Ferrous (magnetic) or electronic implants (due to the magnet in the MRI scanner)
* Claustrophobia

More detailed inclusion/exclusion criteria must be met in order to qualify for the study. The study coordinator will determine eligibility.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers from the community
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Brain connectivity measured by fMRI | One visit

CONTACTS AND LOCATIONS:
Overall Officials: Piero Antuono, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin, United States